CLINICAL TRIAL: NCT07123688
Title: Diagnostic Value of Tc-99mMDP Bone Scan in Assessment of Renal Functions in Cancer Patients Compared to Estimated Glomerular Filtration Rate (eGFR).
Brief Title: Diagnostic Value of Tc-99mMDP Bone Scan in Assessment of Renal Functions in Cancer Patients Compared to Estimated Glomerular Filtration Rate.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Kamel Hamed Ahmed, Resident doctor, Assiut University
Other Study IDs: bone scan in cancer patients
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Cancer Patients Treated by Nephrotoxic Chemotherapy
Keywords: bone scan , renal functions , eGFR

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Tc-99mMDP bone scan — 5 mCi of Tc-99mMDP is used for dynamic renography followed by 15 mCi for post 3-hr whole body imaging.

SUMMARY:
-To compare the glomerular filtration rate obtained by Tc-99mMDP through Gate's method to estimated glomerular filtration rate (eGFR) and assess if we can do metastatic work up and evaluate renal function at a single Tc-99mMDP study, thereby reducing cost, time and radiation exposure.

DETAILED DESCRIPTION:
* Bone scan is one of the frequently used imaging tests in nuclear medicine. It is applied as a test for some oncologic and non-oncologic diseases; the common use is for the detection of bone metastasis from malignant tumors. Renal function may worsen with increasing age, co-morbidities like diabetes, hypertension, acute loss of weight and muscle mass, dehydration and long term use of non-steroidal inflammatory drugs and after some malignancies like multiple myeloma. Therefore renal function assessment is important and can be done by glomerular filtration rate using dGFR. Such a method uses technetium-99m-diethyl-triamine-penta-acetic acid (99mTc-DTPA). Other methods are SCR levels and estimated glomerular filtration rate (eGFR). The use of nephrotoxic drugs such as cisplatin is one of the chemotherapeutic agents in the treatment of a variety of solid tumors; however, it has a side effect of nephrotoxicity. In addition, methotrexate is primarily excreted by the kidneys and estimate of renal function is essential before the use of high-dose therapy.
* Glomerular filtration rate indicates creatinine clearance (CrCl), i.e., a ratio of the concentration of creatinine in serum and urine. Serum creatinine and CrCl have the leading role in the early diagnosis, monitoring and classification of chronic renal insufficiency. MDRD equation may be used for the estimation of glomerular filtration rate, which is accepted due to its simplicity, economic viability and acceptable performance. The most commonly used formula is the "4-varibale MDRD," which estimates GFR using four variables: Serum creatinine, age, race and gender.
* Information about the kidneys can be obtained from bone scan because Tc-99mMDP is excreted through the kidneys. Tc-99mMDP can be an alternative to Tc-99mDTPA for evaluating renal function while conducting bone metastases surveys in patients with urinary tract malignancy with reduced cost and radiation exposure.
* The study aims to investigate the use of Tc-99mMDP for assessing glomerular filtration rate to assess metastatic work up and renal function at a single Tc-99mMDP study, thereby reducing cost, time and radiation exposure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a known history of malignancy treated by nephrotoxic chemotherapy as Cisplatin, who are referred to do bone scan as a part of the metastatic workup. These patients must have recent renal function including serum creatinine, in order to calculate estimated glomerular filtration rate (eGFR) (no chemotherapy is given after the recorded renal function). History of renal problems, previous surgery or medical treatment for the kidney will be reported. Type, duration and dose of chemotherapy also will be reported.

Exclusion Criteria:•

* Patients with known renal failure,Patients refuse to do the scan,Patients with relative or absolute contraindications to do the scan (eg. pregnancy).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with a known history of malignancy treated by nephrotoxic chemotherapy who are referred to do bone scan as a part of the metastatic workup.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Compare the glomerular filtration rate obtained by Tc-99mMDP through Gate's method to estimated glomerular filtration rate in cancer patients treated by nephrotoxic drugs. | from 1 /10/2025 to 1/10/2027
  Compare the glomerular filtration rate obtained by Tc-99mMDP through Gate's method to estimated glomerular filtration rate (eGFR) in adult patients with a known history of malignancy treated by nephrotoxic chemotherapy as Cisplatin, who are referred to do bone scan as a part of the metastatic workup, to evaluate renal function at a single Tc-99mMDP study, thereby reducing cost, time and radiation exposure

REFERENCES:
- [Background] Alqahtani MM. Cisplatin-Induced Renal Failure Measured by Glomerular Filtration Rate (GFR) with 99mTc-DTPA Scans in Cancer Patients: A Systematic Review and Meta-Analysis. Diagnostics (Basel). 2024 Nov 5;14(22):2468. doi: 10.3390/diagnostics14222468. PMID 39594134
- [Background] Javaid A, Munir I, Jaffri SA, Qazi MH, Nawaz MK. A comparison between estimates of glomerular filtration rate using technetium-99m-diethylene-triamine-pentaacetic acid clearance and modification of diet in renal disease equation. Saudi Journal of Medicine & Medical Sciences. 2014;2(3):157-61.
- [Background] Badawy AM, El-Sayed ND, Mohamed OA, Nassar SA, Osman MO. The value of Tc-99mMDP bone scan in assessment of renal functions in urinary tract neoplasm patients after chemotherapy compared toTc-99mDTPA renal scan. Egyptian Journal Nuclear Medicine. 2024;29(2):61-9
- [Background] Krasnow AZ, Hellman RS, Timins ME, Collier BD, Anderson T, Isitman AT. Diagnostic bone scanning in oncology. Semin Nucl Med. 1997 Apr;27(2):107-41. doi: 10.1016/s0001-2998(97)80043-8. PMID 9144855